CLINICAL TRIAL: NCT01865097
Title: Pilot Study of Relaxation Guided Imagery for Treatment of Pain in Parkinson's Disease
Brief Title: Relaxation Guided Imagery for Treatment of Pain in Parkinson's Disease
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Dr. Ilana Schlesinger, Director, Movement Disorders Center, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0494-12
Record Dates: First submitted 2013-05-19; First posted 2013-05-30 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Parkinson's Disease
Keywords: Imagery; Pain; Depression; Non-Motor
MeSH Terms: conditions — Parkinson Disease; Pain; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Relaxation guided imagery (Experimental)
  Interventions: Behavioral: Relaxation guided imagery
- Relaxing music (Active Comparator)
  Interventions: Behavioral: Relaxing music

INTERVENTIONS:
Behavioral: Relaxation guided imagery — An individualized relaxation guided imagery session will be conducted. After the session patients will be given a CD with the relaxation guided imagery and asked to listen to it at home.
  Arms: Relaxation guided imagery
Behavioral: Relaxing music — An individualized session of listening to relaxing music will be conducted. After the session patients will be given a CD with the relaxing music and asked to listen to it at home.
  Arms: Relaxing music

SUMMARY:
Parkinson's disease patients may have severe non-motor symptoms. A common and troublesome non-motor symptom is pain. Currently these symptoms are treated with medication with limited success. Our study aims to determine whether relaxation guided imagery can alleviate pain in Parkinson's disease patients.

DETAILED DESCRIPTION:
Parkinson's disease patients with severe pain without dementia will participate in this study aimed to examine a possible beneficial effect of relaxation guided imagery on pain. This will be a phase I, controlled, single blind and randomized efficacy study in 2 parallel groups. The study will include a baseline assessment of pain severity where after the intervention group will undergo relaxation guided imagery and the control group will listen to relaxing music. After these relaxation session patients will receive a CD with either relaxation guided imagery or relaxing music to listen to at home. Pain severity will be recorded for the following 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic Parkinson's disease suffering from significant pain.

Exclusion Criteria:

* Dementia
* Hearing impairment

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Pain scores on the visual analog scale | 6 weeks
  Numeric rating scale after relaxation guided imagery as compared with baseline

SECONDARY OUTCOMES:
The brief Pain Inventory | 6 weeks
  The brief Pain Inventory after relaxation guided imagery as compared with baseline

OTHER OUTCOMES:
Health status measured by Parkinson's Disease Questionnaire 39(PDQ39) | 6 weeks
  PDQ39 after relaxation guided imagery as compared with baseline
Depression scores on Beck Depression Inventory (BDI) | 6 weeeks
  BDI after relaxation guided imagery as compared with baseline
Non-motor symptom screening questionaire | 6 weeks
  Non-motor symptom screening questionaire after relaxation guided imagery as compared with baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ilana Schlesinger, M.D., Principal Investigator — Rambam Health Care Campus, Haifa, Israel